CLINICAL TRIAL: NCT05959304
Title: A Prospective, Multi-center, Open-label, Phase IV Study to Evaluate the Safety and Effectiveness of Intravitreal Injections (IVI) of Brolucizumab in Patients With Diabetic Macular Edema (DME).
Brief Title: Post Marketing Study to Evaluate the Safety and Effectiveness of Brolucizumab in Patients With Diabetic Macular Edema.
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTH258BIN01
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Macular Edema
Keywords: Vision Loss; Macular Edema; Metamorphopsia
MeSH Terms: conditions — Vision Disorders; Macular Edema | interventions — brolucizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- brolucizumab 6 mg (Experimental): brolucizumab 6 mg intravitreal injection
  Interventions: Drug: brolucizumab

INTERVENTIONS:
Drug: brolucizumab — There is no treatment allocation. Treatment with brolucizumab 6 mg intravitreal injection will be based on the local label/clinical practice.

SUMMARY:
The purpose of this study is to generate additional safety and effectiveness data in Indian Diabetic macular edema (DME) patients that more closely resemble the real-world population intended to be treated with Brolucizumab. This study is being conducted as part of the post-marketing regulatory commitment to the Indian Health authority.

DETAILED DESCRIPTION:
This study is a prospective, non-interventional, open-label, single-arm, multi-center phase IV study to evaluate safety and effectiveness of intravitreal injections (IVI) of brolucizumab in patients with diabetic macular edema (DME) for whom a decision has already been made to be treated with brolucizumab, irrespective of the trial participation. The study period for each patient will be 40 weeks from the informed consent and enrolment in the study.

Assessments/investigations shall be performed in accordance to the local clinical practice and the Investigator's assessed response will be collected in the database. Any patient who suffers from intraocular inflammation (IOI) during the study, treatment with brolucizumab will be discontinued.

Data originating from assessments and evaluations performed at routine patient visits will be collected from the patient's medical records at Baseline, i.e., the start of brolucizumab treatment, and approximately at Week 6, Week 12, Week 18, Week 24, Week 32, Week 36, and at Week 40. Safety data (AEs and SAEs) from any time point during the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥ 18 years old with visual impairment due to DME involving the center of the macula.
2. Patients with type 1 or type 2 diabetes mellitus.
3. Patient or legally acceptable representative (LAR) must provide signed informed consent for participation in the study.

   -

Exclusion Criteria:

1. Concomitant conditions or ocular disorders in the study eye at screening or Baseline which could, in the opinion of the Investigator, prevent response to study treatment or may confound interpretation of study results, compromise visual acuity or require medical or surgical intervention during the study period (e.g., cataract, vitreous hemorrhage, retinal vascular occlusion, retinal detachment, macular hole, or choroidal neovascularization of any cause).
2. Patient with existing or suspected ocular or periocular infection in the study eye.
3. Patient with an existing intraocular inflammation (IOI) in the study eye.
4. Patient who has undergone intraocular surgery including laser photocoagulation in the study eye within 3 months prior to enrollment in this study.
5. Patient with uncontrolled glaucoma defined as intraocular pressure > 25 mmHg despite treatment with anti-glaucoma medication, or according to Investigator's judgment.
6. Patient having scar, fibrosis, and atrophy involving the center of the fovea in the study eye.
7. Active proliferative diabetic retinopathy in the study eye as per Investigator.
8. Patient having history of cardiac or cerebral ischemia in last 6 months prior to enrollment in this study.
9. Previous treatment with any anti-VEGF drugs, steroids (dexamethasone intravitreal implant or triamcinolone acetonide) or other investigational drugs in the study eye.
10. Pregnant or nursing (lactating) women at screening, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG pregnancy test.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence and characteristics of treatment-emergent adverse events during the 40 weeks of treatment with Brolucizumab. | 40 weeks
  To evaluate ocular & non-ocular safety of intravitreal brolucizumab in real-world patients with Diabetic Macular Edema (DME).

SECONDARY OUTCOMES:
Mean change in BCVA from Baseline to Week 40 as measured by ETDRS letters. | Baseline, week 40
  To evaluate the effectiveness of brolucizumab in the management of DME in terms of change in best-corrected visual acuity (BCVA) from Baseline to Week 40 as measured by Early Treatment Diabetic Retinopathy Study (ETDRS) letters.
  Min and max possible scores are 0-100 letters read respectively. A higher score represents better visual functioning.
Percentage of patients with presence/absence of IRF and SRF at Week 40 compared to Baseline. | Baseline, week 40
  To evaluate the effectiveness of brolucizumab on fluid [intraretinal fluid (IRF) and subretinal fluid (SRF)] from Baseline to Week 40.
Mean change in CRT as assessed by Optical Coherence Tomography (OCT) from Baseline to Week 40. | Baseline, week 40
  To evaluate the effectiveness of brolucizumab on central retinal thickness (CRT) from Baseline to Week 40.
Number of brolucizumab injections administered to the patients during 40 weeks of treatment with brolucizumab. | 40 weeks
  To characterize the number of anti-VEGF injections during the 40 weeks of treatment with brolucizumab in the study.
Number of non-injection visits during 40 weeks of treatment with brolucizumab. | 40 weeks
  To characterize the number of non-injection visits during the 40 weeks of treatment with brolucizumab in the study.
Total number of visits during 40 weeks of treatment with brolucizumab. | 40 weeks
  To characterize the total number of visits during the 40 weeks of treatment with brolucizumab in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- India (8):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Coimbatore
  - Novartis Investigative Site, Kolkata
  - Novartis Investigative Site, New Delhi

IPD SHARING:
Plan to Share IPD: No